CLINICAL TRIAL: NCT06156397
Title: The Effect of Technological Based Rehabilitation Practices on Functional Parameters After Breast Cancer Surgery
Brief Title: The Effect of Technological Based Rehabilitation Practices After Breast Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Begüm Büyükerik, Student, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEDU-FTR-BB-001
Record Dates: First submitted 2023-11-25; First posted 2023-12-05 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: rehabilitation; physical therapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Three groups with a conventional therapy control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Physiotherapy Exercise Group (Active Comparator): The exercise protocol will transition from simple to difficult as a result of literature research, and a standard exercise program will be applied, each session lasting 45 minutes.
  Interventions: Other: Standard Physiotherapy Exercise Group
- Telerehabilitation Based Supervised Exercise Group (Active Comparator): Telerehabilitation exercise protocol exercises will last 45 minutes in total, transitioning from simple to difficult, and will be implemented with patients via Zoom.
  Interventions: Other: Telerehabilitation Based Supervised Exercise Group
- Mobile Application Supported Exercise Group (Active Comparator): In the Mobile Application-Based exercise group, a virtual clinic will be created for the patients through the Becure application, and the patients will apply a gradual exercise program that will last approximately 45 minutes, determined by the physiotherapist, and the patients will be followed for 6 weeks through this application.
  Interventions: Other: Mobile Application Supported Exercise Group

INTERVENTIONS:
Other: Standard Physiotherapy Exercise Group — At the beginning of the treatment, breathing exercises, upper extremity pumping exercises, scar tissue massage and flexion movements up to 90 degrees will be applied for the first 2 weeks. 2-6. Between weeks, pendulum exercise, shoulder rotation, lifting overhead with clasped hands while sitting and lying down, wand exercise, snow angels, clock on the wall exercise, m. Pectoralis minor and major stretching, standing trunk rotation, and scapulo-thoracic joint stabilization exercises will be applied. 6-8. In the following weeks, in addition to the previous exercises, strengthening exercises will be applied in all directions with theraband and weights. Exercises will start with 2 sets of 5-10 repetitions and progress to 10-15 repetitions. Exercises will be performed for 45 minutes, twice a week, for a total of 12 sessions, for a total of 6 weeks.
  Arms: Standard Physiotherapy Exercise Group
Other: Telerehabilitation Based Supervised Exercise Group — Exercises will be performed for 45 minutes, twice a week, for a total of 12 sessions, for a total of 6 weeks. In the telerehabilitation group, breathing exercises, upper extremity pumping exercises, scar tissue massage and flexion movements up to 90 degrees will be applied for the first 2 weeks at the beginning of the treatment, through a meeting with the patients via zoom application. 2-6. Between weeks, pendulum exercise, shoulder rotation, lifting overhead with clasped hands while sitting and lying down, wand exercise, snow angels, clock on the wall exercise, m. Pectoralis minor and major stretching, standing trunk rotation, and scapulo-thoracic joint stabilization exercises will be applied. 6-8. In the following weeks, in addition to the previous exercises, strengthening exercises will be applied in all directions with theraband and weights.
  Arms: Telerehabilitation Based Supervised Exercise Group
Other: Mobile Application Supported Exercise Group — With the videos uploaded to the Becure application, breathing exercises, upper extremity pumping exercises, scar tissue massage and flexion movements up to 90 degrees will be applied in the first 2 weeks. 2-6. Between weeks, pendulum exercise, shoulder rotation, lifting overhead with clasped hands while sitting and lying down, wand exercise, snow angels, clock on the wall exercise, m. Pectoralis minor and major stretching, standing trunk rotation, and scapulo-thoracic joint stabilization exercises will be applied. 6-8. Between weeks, in addition to the previous exercises, strengthening exercises will be applied in all directions with theraband and weight. Exercises will start with 2 sets of 5-10 repetitions and progress to 10-15 repetitions.
  Arms: Mobile Application Supported Exercise Group

SUMMARY:
The aim is to investigate the effects of supervised exercise program, telerehabilitation program and mobile application supported exercise program, applied in the acute period after breast cancer surgery, on upper extremity dysfunction.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women. According to the World Health Organization's 2018 data, 11.6% of new cancers worldwide are breast cancer. The overall 5-year survival rates of stage I, II, and III patients are 98%, 92%, and 75%, respectively. Therefore, the survival rate is increasing due to developments in cancer treatment.

The incidence of shoulder mobility impairment after breast cancer surgery was 2% ~ 51%. Postoperative patients' failure to exercise due to fear of pain and affected wound healing leads to poor activity of the upper extremity and shoulder joints, which often leads to limited activity and dysfunction in the affected extremities.

The use of technology in rehabilitation is rapidly increasing, and new technologies provide more motivational participation of patients in their usual care and standard programs. It has been reported that in the acute period after mastectomy, shoulder pain, fatigue, decreased joint range of motion and muscle strength, neuropathy, and consequent limitation of daily living activities.

It has been proven that passive mobilization, general exercise, manual stretching and traditional physiotherapy practices combining them are effective in treating upper extremity pain and restoring functionality after surgery.

There is no study in the literature investigating the effect of an application-based physiotherapy program on upper extremity dysfunction in patients undergoing breast cancer surgery. The aim of this study is to investigate the effects of supervised exercise program, telerehabilitation program and mobile application supported exercise program, applied in the acute period after breast cancer surgery, on upper extremity dysfunction.

Patients who underwent surgery and axillary lymph node dissection will participate in the study. The cases will be randomly divided into three groups. Conventional upper extremity exercises will be planned for the cases in Group 1, telerehabilitation based supervised exercise will be planned for the cases in Group 2, and mobile application-supported exercise treatment will be planned for the cases in Group 3.

In all groups, exercise side effects such as pain, discomfort, and lymphedema development will be monitored by the physiotherapist, with a weekly face to face meeting with the standard physiotherapy exercise group, and with a phone call every 7-10 days with the telerehabilitation and mobile application supported exercise group. Patients who experience adverse effects during or after treatment will be recorded and necessary precautions will be taken.

Treatment program; It will be carried out twice a week for 6 weeks. Each session is scheduled to be approximately 40-45 minutes. Evaluations will be made before and after the application.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with breast cancer and undergoing surgery and having axillary lymph node dissection performed during surgery
* Finding the cases in the post-operative (post-op) 2nd week
* Age range between 30 and 65 years
* Limited shoulder ROM in preoperative evaluations absence
* No speech or hearing problems
* Patients included in the study are volunteers

Exclusion Criteria:

* Previous ipsilateral or contralateral breast cancer surgery
* Presence of active or metastatic cancer focus
* A neurological disease that affects upper extremity functionality or
* Finding orthopedic surgery
* Having hearing or visual impairment
* Carrying a pacemaker
* Presence of infection and open wound
* Finding a drain after surgery
* Cases with mental and cooperation problems

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Baseline Digital Goniometer | six weeks
  The initial and final shoulder range of motion (ROM) of the patients will be recorded in degrees using a digital goniometer. Shoulder ROM measurements will be measured bilaterally and using a standardized protocol.

SECONDARY OUTCOMES:
Disability of Arm, Shoulder and Hand Questionnaire (DASH) | six weeks
  The Injuries to the Arm, Shoulder, and Hand (DASH) questionnaire was developed by the American Academy of Orthopedic Surgeons to assess upper extremity disability and symptoms. The DASH survey consists of three parts. The first part consists of 30 questions that determine the patient's function - symptom score. The first 21 of these questions evaluate the difficulty the patient experiences in performing daily life activities, 5 questions evaluate upper extremity symptoms (pain, pain that occurs with activity, tingling, weakness and difficulty in movement), and the remaining questions evaluate sleep, work, the patient's self-confidence and social life.
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) | six weeks
  The scale is grouped under three subheadings containing 30 questions. Sub-beliefs are the general well-being scale, the functional scale including the subheadings of physical function, general function, cognitive function, mental function and social function, and the symptom consisting of fatigue, pain, stomach brain - enthusiasm, dyspnea, insomnia, fatigue, constipation, diarrhea and material. It includes the scale. The first 28 of the 30 questions in the scale are a four-point Likert type scale and the items are; It is evaluated as Not at all: 1, A little: 2, Quite a bit: 3 or A lot: 4 points. In the 29th and 30th questions of the scale, the patient can be assigned a scale from 1 to 7 (1: Very poor and 7: Excellent), and in the 30th question, a general quality of life evaluation is requested. All scales are scored between 0-100. A high score from the functional scale section indicates good functional status, while a high score from the symptom scale section indicates low vitality.
Muscle Strength Assessment | six weeks
  The upper extremity muscle strength of the subjects will be measured with the J Tech Commander Muscle Tester® manual dynamometer during maximal voluntary isometric muscle contraction. Measurements will be made on the affected and healthy side upper extremities, shoulder flexion and abduction muscle strength in the sitting position, and internal and external rotation muscle strength in the supine position.
  Hand grip strength was evaluated with the Saehan Hydraulic Hand Dynamometer. Measurements will be made on the affected side in a sitting position as defined by the American Society of Hand Therapists, shoulder adducted, arm next to the body, elbow 90° flexed, forearm and wrist in neutral position. The results will be recorded in kg and each measurement will be repeated three times. For result measurements, the values will be averaged and a one-minute rest period will be given between measurements.
Tampa Kinesiophobia Scale (TKS) | six weeks
  Individuals' fear of movement levels will be evaluated using the Tampa Kinesiophobia Scale (TKS). TKS is a checklist consisting of 17 questions and was developed to measure fear of movement/re-injury. The scale evaluates fear of movement with a 4-point Likert-type scoring system (1 = I strongly disagree, 4 = I completely agree). 4,8,12,16. While the total score calculated by reversing the questions is determined between 17-68, a higher score means that the person has a greater fear of movement.
Visual Analog Scale (VAS) | six weeks
  VAS is one of the simple and common methods used to evaluate pain intensity. It is a 10 cm long ruler and generally does not have any markings, numbers or writings on it. Patients are asked to mark the appropriate range for their pain at rest and during activity on a 10 cm long chart (0: no pain; 10 is unbearable pain). The point marked by the patients is measured and recorded in millimeters from the left end with the help of a ruler. It is included in the literature as a sensitive and reliable method.
The Global Rating of Change (GRoC) | six weeks
  The Global Rating of Change (GRoC) is a scale that assesses whether the patient condition has gotten worse, better, or stayed the same and to quantify the magnitude of that change, typically following treatment.
The Functional Assessment of Cancer Therapy - Breast (FACT-B) | six weeks
  The Functional Assessment of Cancer Therapy - Breast (FACT-B) is a 37-item instrument designed to measure five domains of HRQOL in breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Begüm Büyükerik, Principal Investigator — Medipol University
Locations (1):
- The University of Health Sciences Haydarpaşa Numune Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No